CLINICAL TRIAL: NCT05867498
Title: Concurrent and Aerobic Exercise Programs Based on the Polarized Training Intensity Distribution Model on Maximal Oxygen Consumption, Strength, and Body Composition in Overweight and Obese Adults: a Randomized Controlled Trial
Brief Title: Effect of Concurrent and Aerobic Exercise on VO2max, Strength, and Body Composition in Overweight and Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Victor Hugo Arboleda Serna, Dr. Víctor Hugo Arboleda-Serna, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT-AE AFIS-UdeA
Record Dates: First submitted 2023-05-02; First posted 2023-05-22 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers
Keywords: Obesity; Concurrent exercise; Combined training; Circuit-Based Exercise; Cardiorespiratory fitness; Muscle Strength; Body Composition
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concurrent exercise (Experimental): Strength component (circuit-based exercise) 7 exercises:
  * General (2 sets of 15-18 Rep, OMNI-Resistance Exercise Scale 4-5, x 10 s) 180 s
  * Block (3 sets of 12-15 Rep, OMNI-Resistance Exercise Scale 5-6, x 10 s) 70 s
  * Concentrated (3 sets of 10-12 Rep, OMNI-Resistance Exercise Scale 7-8, x 15 s) 110 s
  Aerobic component
  * Low-to-moderate-intensity continuous training: 16 min to 18 min (< VT 1)
  * Interval training: in a block (> VT 2)
    * 5 bouts of 30 s loads. Work:rest ratio: 1:1
    * 4 bouts of 45 s loads. Work:rest ratio: 1:1
    * 5 bouts of 50 s loads. Work:rest ratio: 2:1
    * 4 bouts of 60 s loads. Work:rest ratio: 2:1
    * 3 bouts of 70 s loads. Work:rest ratio: 2:1
    * 4 bouts of 80 s loads. Work:rest ratio: 2:1
  Interventions: Behavioral: Concurrent exercise
- Aerobic exercise (Active Comparator): * Low-to-moderate-intensity continuous training: 36 min (< VT 1)
  * Interval training: in two blocks (> VT 2) 5 bouts of 35 s loads. Work:rest ratio: 1:1 4 bouts of 45 s loads. Work:rest ratio: 1:1 4 bouts of 60 s loads. Work:rest ratio: 2:1 3 bouts of 75 s loads. Work:rest ratio: 2:1 4 bouts of 80 s loads. Work:rest ratio: 2:1
  Interventions: Behavioral: Aerobic exercise

INTERVENTIONS:
Behavioral: Concurrent exercise — Strength component (circuit-based exercise) and aerobic component (based on musicalized and outdoor activities).
  Arms: Concurrent exercise
Behavioral: Aerobic exercise — Low-to-moderate-intensity continuous training and interval training based on musicalized and outdoor activities.
  Arms: Aerobic exercise

SUMMARY:
Concurrent and aerobic physical exercise are recognized strategies for the treatment of overweight and obesity. The interventions of these modalities have been performed with cardiovascular machines or guided execution in their majority, making it possible to improve the health of this population; however, the studies have used high-cost equipment that is not very accessible to the general population. For this reason, we propose to compare the effects of two 12-week programs: concurrent vs. aerobic, using an innovative methodology with musicalized and outdoor activities, little approached by research. The polarized training intensity distribution model, usually used in sports and now applied to physical activity to improve VO2max, muscular strength, and body composition, will be used to determine which intervention is superior in improving these variables.

DETAILED DESCRIPTION:
Twenty-eight people (women and men) will be randomly assigned to a concurrent exercise group (intervention group) and an aerobic exercise group (comparator group), with fourteen people per group. These interventions will be performed for 12 weeks, 3 times per week, with a duration of 60 minutes per session. The first 8 minutes will be of general and specific joint mobility preparing the participants for the central part which will be 47 minutes, and will end with 5 minutes of return to calm.

The concurrent exercise group sessions will have two components, lasting 47 minutes. One of them will be strength exercises with a time of 23 minutes, to perform 7 exercises. In the first four weeks, it will be a general circuit, composed of 2 sets, 15 to 18 repetitions, for 60 seconds, with micro-pauses of 10 seconds between exercises, and 3 minutes between sets. In weeks 5 to 8, it will be a block circuit, consisting of 3 sets, 12 to 15 repetitions, for 45 seconds, with micro-pauses of 10 seconds between exercises and 70 seconds between sets. For weeks 9 to 12, it will be a concentrated circuit, consisting of 3 sets, 8 to 12 repetitions, for 35 seconds, with micro-pauses of 15 seconds between exercises and 110 seconds between sets.

The aerobic component will have a duration equal to the strength component (24 minutes). A variable continuous method will be applied for the first 18 minutes through rumba-aerobic (ballroom and folkloric dance steps), at an intensity lower than the ventilatory threshold 1 (VT 1). For the remaining 6 minutes, an intervallic method will be used at an intensity > VT 2, with combat gestures (fists, knees, and plantar flexions). Progression of the loads during the 12 weeks of intervention: Weeks 1 and 2: 5 loads of 30 seconds and 30 seconds of recovery.

Weeks 3 and 4: 4 loads of 45 seconds and 45 seconds of recovery. Weeks 5 to 7: 5 loads of 50 seconds and 25 seconds of recovery. Week 8: 4 loads of 60 seconds and 30 seconds of recovery. Weeks 9 to 11: 3 loads of 70 seconds and 35 seconds of recovery. Week 12: 4 loads of 80 and 40 seconds of recovery.

The aerobic group, will perform the same methods, rumba steps, combat gestures, intensities, and time of the central part of the aerobic component of the concurrent exercise group, but will be differentiated by performing in the continuous method for a duration of 36 minutes and in the interval method will have the following progression:

Weeks 1 and 2: 2 blocks by 5 loads of 35 seconds and 35 seconds of recovery. Weeks 3 and 4: 2 blocks by 4 loads of 45 seconds and 45 seconds of recovery. Weeks 5 to 8: 2 blocks by 4 loads of 60 seconds and 30 seconds of recovery. Weeks 9 to 11: 2 blocks by 3 loads of 75 seconds and 37.5 seconds of recovery. Week 12: 2 blocks by 4 loads of 80 seconds and 40 seconds of recovery.

All participants will have their maximal oxygen consumption, muscle strength, and body composition evaluated before the beginning of week 1 and at the end of week 12.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 59 years old.
* BMI >25.0.
* Waist circumference ≥85cm in women, and ≥94cm in men.
* Individuals participating voluntarily.

Exclusion Criteria:

* History of cardiovascular and pulmonary disease.
* Uncontrolled psychiatric problems.
* People under treatment with anticoagulants, beta-blockers, calcium antagonists, and bronchodilators.
* Having osteo-muscular problems that may affect participation in exercise sessions.
* Pregnant women.
* People with a nutritional plan for weight loss.
* Smokers.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Change in maximal oxygen consumption | Baseline and 12-weeks
  A graded exercise test on a cycle ergometer (ERGO-FIT, Germany) will obtain maximal oxygen consumption (VO2max) using a METAMAX 3B gas analyzer (CORTEX, Germany). VO2max will be reported in ml/kg/min.

SECONDARY OUTCOMES:
Change in mean propulsive velocity | Baseline and 12-weeks
  Mean propulsive velocity (m/s), will be assessed by a progressive half squat test on a Smith machine, with a T-Force System linear encoder (ERGOTECH, Spain).
Change in maximum velocity | Baseline and 12-weeks
  Maximum velocity (m/s), will be assessed by a progressive half squat test on a Smith machine, with a T-Force System linear encoder (ERGOTECH, Spain).
Change in peak maximum power | Baseline and 12-weeks
  Peak maximum power (W), will be assessed by a progressive half squat test on a Smith machine, with a T-Force System linear encoder (ERGOTECH, Spain).
Change in body fat | Baseline and 12-weeks
  Body fat (%), will be obtained using an InBody 270 body composition analyzer (InBody, USA).
Change in muscle mass | Baseline and 12-weeks
  Muscle mass (kg), will be obtained using an InBody 270 body composition analyzer (InBody, USA).
Change in visceral fat level | Baseline and 12-weeks
  Visceral fat level (>10 high, <10 low), will be obtained using an InBody 270 body composition analyzer (InBody, USA).
Change in body weight | Baseline and 12-weeks
  Body weight (kg), will be obtained using an InBody 270 body composition analyzer (InBody, USA).
Change in waist circumference | Baseline and 12-weeks
  Waist circumference (cm), will be obtained using a tape measure (SECA).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Antioquia, Medellín, Antioquia, Colombia